CLINICAL TRIAL: NCT03671785
Title: A Prospective, Randomized, Placebo-Controlled Pilot Study to Characterize the Intestinal Microbiome and to Evaluate the Safety and Fecal Microbiome Changes Following Twice Weekly Administration of Lyophilized PRIM-DJ2727 or Placebo Given Orally for 12 Weeks in Subjects With Parkinson's Disease
Brief Title: Study of the Fecal Microbiome in Patients With Parkinson's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Kelsey Research Foundation (Other)
Responsible Party: Principal Investigator, Herbert DuPont, MD, Professor of Infectious Diseases, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSC-SPH-18-0621
Record Dates: First submitted 2018-09-12; First posted 2018-09-14 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active group treated with healthy fecal microbiota (Experimental)
  Interventions: Drug: PRIM-DJ2727
- Placebo group (Experimental)
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: PRIM-DJ2727 — Twice filtered fecal microbiota product from three screened healthy donors will be lyophilized and encapsulated in enteric-coated capsules. Each dose of enteric coated capsules consists of 60 grams of stool and will be administered orally twice-weekly for 12 consecutive weeks
  Arms: Active group treated with healthy fecal microbiota
Drug: Placebo oral capsule — Placebo capsule will be identical to PRIM-DJ2727 but will not contain intestinal bacteria. The placebo will consist of Lactose (spray-dried United States Pharmacopeia (USP) 64.385gm), food color, powdered Black, Brown, and Yellow in the enteric capsules. Placebo will be administered orally twice-weekly for 12 consecutive weeks
  Arms: Placebo group

SUMMARY:
The purpose of this study is to characterize the intestinal microbiome in subjects with Parkinson's disease and to determine safety and trends in improvements in diversity of colonic microbiome following administration of lyophilized PRIM-DJ2727

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of Parkinson's Disease (PD) for less than or equal to 10 years based on the United Kingdom Brain Bank Criteria and the Modified Hoehn-Yahr (H&Y) staging system of less than 3 in the "OFF medicine" state of at least 8-12 hours (subjects should have an asymmetric and unilateral symptoms onset).
* Mild microsomia to anosmia (The University of Pennsylvania Smell Identification Test (UPSIT) less than 33), which is supportive of idiopathic PD.
* Robust response to dopaminergic therapy (defined as greater than 33% reduction in symptoms (on the Unified Parkinson's Disease Rating Scale part III (UPDRS-III)) when measured in the ON medicine state compared to OFF state.
* Subject has a history of constipation.
* Sexually active male and female subjects of child-bearing potential agree to use an effective method of birth control during the study.
* Female subjects of child-bearing potential must have a negative urine Qualitative Human chorionic gonadotropin (hCG) pregnancy test at enrollment and on the Week 1, Day 1 of the Treatment prior to administration of study drug.
* Willing and able to sign an informed consent form and attend study assessments and follow ups.
* Subject has an attending physician who will provide non-transplant care for the subject.
* Subject is able to maintain a stable Parkinson's therapy medical regimen during participation in the study.

Exclusion Criteria:

* Unable to take multiple capsules orally.
* Montreal Cognitive Assessment (MoCA) Score less than or equal to 23.
* Atypical, vascular or drug-induced Parkinsonism.
* Clinical features of psychosis or refractory hallucinations.
* Unstable Parkinson's disease symptomatic therapy (defined as recent changes or additions to the PD regimen).
* Compromised immune system (e.g. primary immune disorders or clinical immunosuppression due to a medical condition or medication e.g. taking systemic steroids greater than 20 milligrams (mg) a day or prednisone-equivalent)
* Receipt of systemic non-topical antibiotic therapy currently or within 14 days of enrollment.
* Prior Deep Brain Stimulation, or surgical intervention for PD, intravenous glutathione therapy or stem cell therapy.
* History of medium or large vessel cerebrovascular accidents.
* History of use of an investigational drug within 90 days prior to the screening visit.
* Positive results for human immunodeficiency virus (HIV) or Hepatitis B / C.
* Current history for active states of Inflammatory bowel disease, Irritable bowel syndrome, microscopic colitis, celiac disease, short gut syndrome, colostomy, colectomy, gastrointestinal fistulae or strictures.
* History of significant uncontrolled systemic disease that in the opinion of the study investigator could interfere with study participation and/or objectives.
* Life expectancy of less than 1 year.
* In the opinion of investigator, subject for any reason, should be excluded from the study

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2022-10-09 (Actual); Study Completion 2022-10-12 (Actual)

PRIMARY OUTCOMES:
Microbiome Diversity in Fecal Samples as Indicated by the Shannon Diversity Index | baseline
  The Shannon diversity index is used to characterize species diversity in a community. Shannon's index accounts for both abundance and evenness of the species present. A high index value would represent a diverse and equally distributed community, and lower values represent a less diverse community. A value of 0 would represent a community with just one species. Typical values are generally between 1.5 and 3.5.
Microbiome Diversity in Fecal Samples as Indicated by the Shannon Diversity Index | week 6
  The Shannon diversity index is used to characterize species diversity in a community. Shannon's index accounts for both abundance and evenness of the species present. A high index value would represent a diverse and equally distributed community, and lower values represent a less diverse community. A value of 0 would represent a community with just one species. Typical values are generally between 1.5 and 3.5.
Microbiome Diversity in Fecal Samples as Indicated by the Shannon Diversity Index | week 13
  The Shannon diversity index is used to characterize species diversity in a community. Shannon's index accounts for both abundance and evenness of the species present. A high index value would represent a diverse and equally distributed community, and lower values represent a less diverse community. A value of 0 would represent a community with just one species. Typical values are generally between 1.5 and 3.5.
Microbiome Diversity in Fecal Samples as Indicated by the Shannon Diversity Index | month 4
  The Shannon diversity index is used to characterize species diversity in a community. Shannon's index accounts for both abundance and evenness of the species present. A high index value would represent a diverse and equally distributed community, and lower values represent a less diverse community. A value of 0 would represent a community with just one species. Typical values are generally between 1.5 and 3.5.
Microbiome Diversity in Fecal Samples as Indicated by the Shannon Diversity Index | month 6
  The Shannon diversity index is used to characterize species diversity in a community. Shannon's index accounts for both abundance and evenness of the species present. A high index value would represent a diverse and equally distributed community, and lower values represent a less diverse community. A value of 0 would represent a community with just one species. Typical values are generally between 1.5 and 3.5.
Microbiome Diversity in Fecal Samples as Indicated by the Shannon Diversity Index | month 9
  The Shannon diversity index is used to characterize species diversity in a community. Shannon's index accounts for both abundance and evenness of the species present. A high index value would represent a diverse and equally distributed community, and lower values represent a less diverse community. A value of 0 would represent a community with just one species. Typical values are generally between 1.5 and 3.5.
Microbiome Richness in Fecal Samples as Indicated by the Number of Taxonomies per Participant | baseline
Microbiome Richness in Fecal Samples as Indicated by the Number of Taxonomies per Participant | week 6
Microbiome Richness in Fecal Samples as Indicated by the Number of Taxonomies per Participant | week 13
Microbiome Richness in Fecal Samples as Indicated by the Number of Taxonomies per Participant | month 4
Microbiome Richness in Fecal Samples as Indicated by the Number of Taxonomies per Participant | month 6
Microbiome Richness in Fecal Samples as Indicated by the Number of Taxonomies per Participant | month 9
Any untoward medical occurrence after fecal microbiota transplantation (FMT) | 9 months after treatments starts

SECONDARY OUTCOMES:
Number of participants with an increase in flora diversity in fecal samples | 9 months after treatments starts
Change in number of bowel movements per day | Baseline, 2 weeks
  The 2 week data point will be the average of bowel movements per day over the two weeks after initiation of treatment.
Motor function as characterized by Unified Parkinson's Disease Rating Scale (UPDRS) Total Score | baseline
  UPDRS is a disability and impairment scale for PD progression and consists of 4 sections; I: evaluation of mentation, behavior, and mood (13 questions) II: evaluation of activities of daily living including speech, swallowing, handwriting, dressing, hygiene, falling, salivating, turning in bed, walking, and cutting food (13 questions) III: motor examination (33 scores based on 18 questions with right, left or other body distributions scores) IV: motor complications (6 questions)
  All items have 5 response options: 0 = normal, 1 = slight (symptoms/ signs with sufficiently low frequency or intensity to cause no impact on function), 2 = mild (symptoms/ signs of frequency or intensity sufficient to cause a modest impact on function, 3 = moderate (symptoms/ signs sufficiently frequent or intense to impact considerably, but not prevent function), 4 = severe (symptoms/ signs that prevent function).
  Total Score ranges from 0 to 260, with higher scores indicating a worse outcome.
Motor function as characterized by Unified Parkinson's Disease Rating Scale (UPDRS) Total Score | 4 months
  UPDRS is a disability and impairment scale for PD progression and consists of 4 sections; I: evaluation of mentation, behavior, and mood (13 questions) II: evaluation of activities of daily living including speech, swallowing, handwriting, dressing, hygiene, falling, salivating, turning in bed, walking, and cutting food (13 questions) III: motor examination (33 scores based on 18 questions with right, left or other body distributions scores) IV: motor complications (6 questions)
  All items have 5 response options: 0 = normal, 1 = slight (symptoms/ signs with sufficiently low frequency or intensity to cause no impact on function), 2 = mild (symptoms/ signs of frequency or intensity sufficient to cause a modest impact on function, 3 = moderate (symptoms/ signs sufficiently frequent or intense to impact considerably, but not prevent function), 4 = severe (symptoms/ signs that prevent function).
  Total Score ranges from 0 to 260, with higher scores indicating a worse outcome.
Motor function as characterized by Unified Parkinson's Disease Rating Scale (UPDRS) Total Score | 9 months
  UPDRS is a disability and impairment scale for PD progression and consists of 4 sections; I: evaluation of mentation, behavior, and mood (13 questions) II: evaluation of activities of daily living including speech, swallowing, handwriting, dressing, hygiene, falling, salivating, turning in bed, walking, and cutting food (13 questions) III: motor examination (33 scores based on 18 questions with right, left or other body distributions scores) IV: motor complications (6 questions)
  All items have 5 response options: 0 = normal, 1 = slight (symptoms/ signs with sufficiently low frequency or intensity to cause no impact on function), 2 = mild (symptoms/ signs of frequency or intensity sufficient to cause a modest impact on function, 3 = moderate (symptoms/ signs sufficiently frequent or intense to impact considerably, but not prevent function), 4 = severe (symptoms/ signs that prevent function).
  Total Score ranges from 0 to 260, with higher scores indicating a worse outcome.
Motor function as characterized by Unified Parkinson's Disease Rating Scale (UPDRS) Motor Score | baseline
  UPDRS is a disability and impairment scale for PD progression and consists of 4 sections; I: evaluation of mentation, behavior, and mood (13 questions) II: evaluation of activities of daily living including speech, swallowing, handwriting, dressing, hygiene, falling, salivating, turning in bed, walking, and cutting food (13 questions) III: motor examination (33 scores based on 18 questions with right, left or other body distributions scores) IV: motor complications (6 questions)
  All items have 5 response options: 0 = normal, 1 = slight (symptoms/ signs with sufficiently low frequency or intensity to cause no impact on function), 2 = mild (symptoms/ signs of frequency or intensity sufficient to cause a modest impact on function, 3 = moderate (symptoms/ signs sufficiently frequent or intense to impact considerably, but not prevent function), 4 = severe (symptoms/ signs that prevent function).
  Motor Score ranges from 0 to 156, with higher scores indicating a worse outcome.
Motor function as characterized by Unified Parkinson's Disease Rating Scale (UPDRS) Motor Score | 4 months
  UPDRS is a disability and impairment scale for PD progression and consists of 4 sections; I: evaluation of mentation, behavior, and mood (13 questions) II: evaluation of activities of daily living including speech, swallowing, handwriting, dressing, hygiene, falling, salivating, turning in bed, walking, and cutting food (13 questions) III: motor examination (33 scores based on 18 questions with right, left or other body distributions scores) IV: motor complications (6 questions)
  All items have 5 response options: 0 = normal, 1 = slight (symptoms/ signs with sufficiently low frequency or intensity to cause no impact on function), 2 = mild (symptoms/ signs of frequency or intensity sufficient to cause a modest impact on function, 3 = moderate (symptoms/ signs sufficiently frequent or intense to impact considerably, but not prevent function), 4 = severe (symptoms/ signs that prevent function).
  Motor Score ranges from 0 to 156, with higher scores indicating a worse outcome.
Motor function as characterized by Unified Parkinson's Disease Rating Scale (UPDRS) Motor Score | 9 months
  UPDRS is a disability and impairment scale for PD progression and consists of 4 sections; I: evaluation of mentation, behavior, and mood (13 questions) II: evaluation of activities of daily living including speech, swallowing, handwriting, dressing, hygiene, falling, salivating, turning in bed, walking, and cutting food (13 questions) III: motor examination (33 scores based on 18 questions with right, left or other body distributions scores) IV: motor complications (6 questions)
  All items have 5 response options: 0 = normal, 1 = slight (symptoms/ signs with sufficiently low frequency or intensity to cause no impact on function), 2 = mild (symptoms/ signs of frequency or intensity sufficient to cause a modest impact on function, 3 = moderate (symptoms/ signs sufficiently frequent or intense to impact considerably, but not prevent function), 4 = severe (symptoms/ signs that prevent function).
  Motor Score ranges from 0 to 156, with higher scores indicating a worse outcome.
Parkinson's disease symptoms as assessed by the Modified Hoehn and Yahr Scale | baseline
  Modified H&Y scale will be used as a staging instrument to monitor progression of PD's symptoms. It defines broad categories of motor function in PD starting at Stage 0: no signs of disease to the highest stage 5: wheelchair bound or bedridden unless aided.
Parkinson's disease symptoms as assessed by the Modified Hoehn and Yahr Scale | 4 months
  Modified H&Y scale will be used as a staging instrument to monitor progression of PD's symptoms. It defines broad categories of motor function in PD starting at Stage 0: no signs of disease to the highest stage 5: wheelchair bound or bedridden unless aided.
Parkinson's disease symptoms as assessed by the Modified Hoehn and Yahr Scale | 9 months
  Modified H&Y scale will be used as a staging instrument to monitor progression of PD's symptoms. It defines broad categories of motor function in PD starting at Stage 0: no signs of disease to the highest stage 5: wheelchair bound or bedridden unless aided.
Cognitive domains characterized by using Montreal Cognitive Assessment | baseline
  MoCA is a rapid screening instrument for mild cognitive dysfunction. It assess different cognitive domains: attention and concentration, executive functions, memory, language, visuo-constructional skills, conceptual thinking, calculations, and orientation. The total score ranges from 0 to 30; a score of 26 or above is considered normal. MoCA will be performed at the enrollment for baseline and the clinic visit on 9 month for study endpoint assessment, and early termination visit (if applicable).
Cognitive domains characterized by using Montreal Cognitive Assessment | 4 months
  MoCA is a rapid screening instrument for mild cognitive dysfunction. It assess different cognitive domains: attention and concentration, executive functions, memory, language, visuo-constructional skills, conceptual thinking, calculations, and orientation. The total score ranges from 0 to 30; a score of 26 or above is considered normal. MoCA will be performed at the enrollment for baseline and the clinic visit on 9 month for study endpoint assessment, and early termination visit (if applicable).
Cognitive domains characterized by using Montreal Cognitive Assessment | 9 months
  MoCA is a rapid screening instrument for mild cognitive dysfunction. It assess different cognitive domains: attention and concentration, executive functions, memory, language, visuo-constructional skills, conceptual thinking, calculations, and orientation. The total score ranges from 0 to 30; a score of 26 or above is considered normal. MoCA will be performed at the enrollment for baseline and the clinic visit on 9 month for study endpoint assessment, and early termination visit (if applicable).
Change in Sense of Smell as assessed by the University of Pennsylvania Smell Identification Test (UPSIT) | baseline, 9 months
  The UPSIT is a comprehensive 40-item self-administered olfactory test that provides an absolute indication of smell loss (anosmia; mild, moderate or severe microsomia). The range of scores is 0 to 40, and a higher score indicates better olfaction
Qualify of life as assessed by the Parkinson's disease Questionnaire (PDQ-39) | baseline
  The Parkinson's disease Questionnaire (PDQ-39) is a 39 questions self-completed questionnaire that comprises 8 domains: mobility (10 items), activities of daily living (6 items), emotional well-being (6 items), stigma (4 items), social support (3 items), cognition (4 items), communication (3 items) and bodily discomfort (3 items). All items are assumed to impact Quality of Life (QoL) and must be answered to compute scores for each dimension. Questions are answered based on experiences from the preceding month using a 5-point ordinal scoring system: 0 = never, 1 = occasionally, 2 = sometimes, 3 = often, 4 = always. Overall score ranges from 0 = never have difficulty to 100 = always have difficulty. For each of the 8 domains, the domain score is the sum of scores in the domain divided by the maximum possible score of all items in the domain, multiplied by 100. The overall score is the sum of all 8 domain scores divided by 8.
Qualify of life as assessed by the Parkinson's disease Questionnaire (PDQ-39) | 4 months
  The Parkinson's disease Questionnaire (PDQ-39) is a 39 questions self-completed questionnaire that comprises 8 domains: mobility (10 items), activities of daily living (6 items), emotional well-being (6 items), stigma (4 items), social support (3 items), cognition (4 items), communication (3 items) and bodily discomfort (3 items). All items are assumed to impact QoL and must be answered to compute scores for each dimension. Questions are answered based on experiences from the preceding month using a 5-point ordinal scoring system: 0 = never, 1 = occasionally, 2 = sometimes, 3 = often, 4 = always. Overall score ranges from 0 = never have difficulty to 100 = always have difficulty. For each of the 8 domains, the domain score is the sum of scores in the domain divided by the maximum possible score of all items in the domain, multiplied by 100. The overall score is the sum of all 8 domain scores divided by 8.
Qualify of life as assessed by the Parkinson's disease Questionnaire (PDQ-39) | 9 months
  The Parkinson's disease Questionnaire (PDQ-39) is a 39 questions self-completed questionnaire that comprises 8 domains: mobility (10 items), activities of daily living (6 items), emotional well-being (6 items), stigma (4 items), social support (3 items), cognition (4 items), communication (3 items) and bodily discomfort (3 items). All items are assumed to impact QoL and must be answered to compute scores for each dimension. Questions are answered based on experiences from the preceding month using a 5-point ordinal scoring system: 0 = never, 1 = occasionally, 2 = sometimes, 3 = often, 4 = always. Overall score ranges from 0 = never have difficulty to 100 = always have difficulty. For each of the 8 domains, the domain score is the sum of scores in the domain divided by the maximum possible score of all items in the domain, multiplied by 100. The overall score is the sum of all 8 domain scores divided by 8.
Quality of Life as assessed by the Parkinson Disease Non-Motor Symptoms (PD NMS) Questionnaire | baseline
  The range of scores is 0 to 30. A score of under 10 is mild, 10-20 moderate and over 20 severe.
Quality of Life as assessed by the Parkinson Disease Non-Motor Symptoms (PD NMS) Questionnaire | 4 months
  The range of scores is 0 to 30. A score of under 10 is mild, 10-20 moderate and over 20 severe.
Quality of Life as assessed by the Parkinson Disease Non-Motor Symptoms (PD NMS) Questionnaire | 9 months
  The range of scores is 0 to 30. A score of under 10 is mild, 10-20 moderate and over 20 severe.
Number of participants who changed required PD symptomatic therapy after treatment | 9 months after treatment
Number of participants with worsening of PD symptoms or other potential microbial-mediated disorders | 9 months after treatment
Anxiety as assessed by the Parkinson Anxiety Scale (PAS) | baseline
  The Parkinson Anxiety Scale (PAS) is an anxiety measure scale for use in PD patients. This is a 12-item observer or patient-rated scale with three subscales, for persistent and episodic anxiety, and avoidance behavior. Items are scored on a 5-point Likert scale, with '0' meaning 'not or never' and '4' meaning 'severe or almost always'. Total score ranges from 0 to 48, with higher scores indicating worse outcomes.
Anxiety as assessed by the Parkinson Anxiety Scale (PAS) | 4 months
  The Parkinson Anxiety Scale (PAS) is an anxiety measure scale for use in PD patients. This is a 12-item observer or patient-rated scale with three subscales, for persistent and episodic anxiety, and avoidance behavior. Items are scored on a 5-point Likert scale, with '0' meaning 'not or never' and '4' meaning 'severe or almost always'. Total score ranges from 0 to 48, with higher scores indicating worse outcomes.
Anxiety as assessed by the Parkinson Anxiety Scale (PAS) | 9 months
  The Parkinson Anxiety Scale (PAS) is an anxiety measure scale for use in PD patients. This is a 12-item observer or patient-rated scale with three subscales, for persistent and episodic anxiety, and avoidance behavior. Items are scored on a 5-point Likert scale, with '0' meaning 'not or never' and '4' meaning 'severe or almost always'. Total score ranges from 0 to 48, with higher scores indicating worse outcomes.
Depression as assessed by the Geriatric Depression Scale Short form (GDS-SF) | baseline
  The Geriatric Depression Scale Short form (GDS-SF) is 15-item screening tool that is used to identify depression in older adults. The total score is 0 to 15, with a score of 5 or greater suggesting depression.
Depression as assessed by the Geriatric Depression Scale Short form (GDS-SF) | 4 months
  The Geriatric Depression Scale Short form (GDS-SF) is 15-item screening tool that is used to identify depression in older adults.The total score is 0 to 15, with a score of 5 or greater suggesting depression.
Depression as assessed by the Geriatric Depression Scale Short form (GDS-SF) | 9 months
  The Geriatric Depression Scale Short form (GDS-SF) is 15-item screening tool that is used to identify depression in older adults.The total score is 0 to 15, with a score of 5 or greater suggesting depression.
Change in gastric emptying time (GET) as assessed by the Smart Pill® (SP) Wireless pH/pressure recording capsule | baseline, 13 weeks
  Smart Pill will be used to assess gastrointestinal dysmotility in PD patients before and after 12- week treatment. Smart Pill will be administered first during the run-In period clinic visit and again at Week 13 clinic visit following the completion of 12-week treatment. After an overnight fast, subjects will ingest the Smart Pill capsule with a nutrient bar (Smart Bar, 243 kcal) and will be instructed to wear a data receiver for 5 days or until the expulsion of the Smart Pill. After expulsion of the Smart Pill in approximately 5 days, subject will return the data receiver. Data receiver can either be dropped by or mailed via FedEx to the study site. Changes in gastric emptying time (GET), small bowel transit time (SBTT), colon transit time (CTT), small/ large bowel transit time (SLBTT) and whole gut transit time (WGTT) will be assessed by parameters established by the company providing the Smart Pill capsule.
Change in small bowel transit time (SBTT) as assessed by the Smart Pill® (SP) Wireless pH/pressure recording capsule | baseline, 13 weeks
  Smart Pill will be used to assess gastrointestinal dysmotility in PD patients before and after 12- week treatment. Smart Pill will be administered first during the run-In period clinic visit and again at Week 13 clinic visit following the completion of 12-week treatment. After an overnight fast, subjects will ingest the Smart Pill capsule with a nutrient bar (Smart Bar, 243 kcal) and will be instructed to wear a data receiver for 5 days or until the expulsion of the Smart Pill. After expulsion of the Smart Pill in approximately 5 days, subject will return the data receiver. Data receiver can either be dropped by or mailed via FedEx to the study site. Changes in gastric emptying time (GET), small bowel transit time (SBTT), colon transit time (CTT), small/ large bowel transit time (SLBTT) and whole gut transit time (WGTT) will be assessed by parameters established by the company providing the Smart Pill capsule.
Change in colon transit time (CTT) as assessed by the Smart Pill® (SP) Wireless pH/pressure recording capsule | baseline, 13 weeks
  Smart Pill will be used to assess gastrointestinal dysmotility in PD patients before and after 12- week treatment. Smart Pill will be administered first during the run-In period clinic visit and again at Week 13 clinic visit following the completion of 12-week treatment. After an overnight fast, subjects will ingest the Smart Pill capsule with a nutrient bar (Smart Bar, 243 kcal) and will be instructed to wear a data receiver for 5 days or until the expulsion of the Smart Pill. After expulsion of the Smart Pill in approximately 5 days, subject will return the data receiver. Data receiver can either be dropped by or mailed via FedEx to the study site. Changes in gastric emptying time (GET), small bowel transit time (SBTT), colon transit time (CTT), small/ large bowel transit time (SLBTT) and whole gut transit time (WGTT) will be assessed by parameters established by the company providing the Smart Pill capsule.
Change in small/large bowel transit time (SLBTT) as assessed by the Smart Pill® (SP) Wireless pH/pressure recording capsule | baseline, 13 weeks
  Smart Pill will be used to assess gastrointestinal dysmotility in PD patients before and after 12- week treatment. Smart Pill will be administered first during the run-In period clinic visit and again at Week 13 clinic visit following the completion of 12-week treatment. After an overnight fast, subjects will ingest the Smart Pill capsule with a nutrient bar (Smart Bar, 243 kcal) and will be instructed to wear a data receiver for 5 days or until the expulsion of the Smart Pill. After expulsion of the Smart Pill in approximately 5 days, subject will return the data receiver. Data receiver can either be dropped by or mailed via FedEx to the study site. Changes in gastric emptying time (GET), small bowel transit time (SBTT), colon transit time (CTT), small/ large bowel transit time (SLBTT) and whole gut transit time (WGTT) will be assessed by parameters established by the company providing the Smart Pill capsule.
Change in whole gut transit time (WGTT) as assessed by the Smart Pill® (SP) Wireless pH/pressure recording capsule | baseline, 13 weeks
  Smart Pill will be used to assess gastrointestinal dysmotility in PD patients before and after 12- week treatment. Smart Pill will be administered first during the run-In period clinic visit and again at Week 13 clinic visit following the completion of 12-week treatment. After an overnight fast, subjects will ingest the Smart Pill capsule with a nutrient bar (Smart Bar, 243 kcal) and will be instructed to wear a data receiver for 5 days or until the expulsion of the Smart Pill. After expulsion of the Smart Pill in approximately 5 days, subject will return the data receiver. Data receiver can either be dropped by or mailed via FedEx to the study site. Changes in gastric emptying time (GET), small bowel transit time (SBTT), colon transit time (CTT), small/ large bowel transit time (SLBTT) and whole gut transit time (WGTT) will be assessed by parameters established by the company providing the Smart Pill capsule.

CONTACTS AND LOCATIONS:
Overall Officials: Herbert L DuPont, MD, Principal Investigator — University of Texas Health Science Center School of Public Health
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] DuPont HL, Suescun J, Jiang ZD, Brown EL, Essigmann HT, Alexander AS, DuPont AW, Iqbal T, Utay NS, Newmark M, Schiess MC. Fecal microbiota transplantation in Parkinson's disease-A randomized repeat-dose, placebo-controlled clinical pilot study. Front Neurol. 2023 Mar 2;14:1104759. doi: 10.3389/fneur.2023.1104759. eCollection 2023. PMID 36937520